CLINICAL TRIAL: NCT04155281
Title: Consumption of New Psychoactive Substances in Intoxicated Patients During the Winter Activities
Brief Title: New Psychoactive Substances in Intoxicated Patients During the Winter Activities
Acronym: SkiTox
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC19.214; 2019-A02214-53 (Other: ID RCB)
Record Dates: First submitted 2019-09-27; First posted 2019-11-07 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Acute Intoxication; Psychoactive Substance Use
Keywords: Intoxication; Psychoactive Substance ; Ski
MeSH Terms: interventions — Urinalysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- suspicion of intoxication: New Psychoactive Substances research in urine
  Interventions: Other: urine analysis

INTERVENTIONS:
Other: urine analysis — New Psychoactive Substances research in urine at admission in unit care

SUMMARY:
The purpose of this research is to identify the New Psychoactive Substances (NPS) that are responsible for intoxicating patients in ski resort during winter activities.

DETAILED DESCRIPTION:
The New Psychoactive Substances expose to an additional risk of overdose or death due to their potency. These New Psychoactive Substances are used voluntarily by users wishing to test new substances, but also involuntarily because of association (unknowingly users) with more "conventional" drugs such as cocaine or heroin in the self-administered powder. These intoxications are still poorly known and the investigators believe that the identification of New Psychoactive Substances among the drugs consumed, and the association of their consumption with the appearance of a particular symptomatology allow the physician to guide the diagnosis and facilitate the care of future patients.

ELIGIBILITY:
Inclusion Criteria:

* Admission to emergency, resuscitation or intensive care departments involved in the study
* Anamnestic and / or clinical suspicion of acute drug poisoning according to International Classification of Diseases-10 criteria
* Patient coming from a ski resort from the pre-established list
* urine sample available as part of the treatment
* person understanding French or English
* Non-opposition to the study

Exclusion Criteria:

* Suspicion of alcohol intoxication alone
* Suspicion of voluntary drug poisoning
* Suspicion of intentional intoxication by others
* Pregnant or breastfeeding women
* Major mentioned in Articles L1121-6 and 1121-8 of french public health code
* Patients in the exclusion period of another research involving the human person type 1 or 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient will be included at admission to hospital (Grenoble alpes university hospital, CH Albertville-Moûtiers and Centre Hospitalier Métropole Savoie/Chambéry). After collecting his/her non-opposition to the study, the urine sample of the medical care will be kept and send to the central lab for analysis and dentifation of new psychoactive substances.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
positive urinary sample | Day 0
  proportion of urine samples positive for New Psychoactive Substances and related, among patients suspected of intoxication and from a ski resort, in winter.

SECONDARY OUTCOMES:
incidence of toxidromes | baseline
  Clinical symptoms observed in intoxicated patients
polyintoxication frequency | baseline
  Percentage of co-intoxications
morbidity of intoxication | baseline and month 1
  length of stay in hospital
morbidity of intoxication | baseline and month 1
  Percentage of Intensive Care Unit admissions
incidence of intoxication medical care | day 1
  names of therapies implemented within 24 hours of admission

CONTACTS AND LOCATIONS:
Overall Officials: Damien VIGLINO, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (3):
- France (3):
  - Centre Hospitalier Métropole Savoie (Chaméry), Chambéry, Savoie
  - CH Albertville Moutiers, Albertville
  - University Hospital Grenoble, Grenoble

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rivera JV, Vance EG, Rushton WF, Arnold JK. Novel Psychoactive Substances and Trends of Abuse. Crit Care Nurs Q. 2017 Oct/Dec;40(4):374-382. doi: 10.1097/CNQ.0000000000000174. PMID 28834859
- [Background] Yang F-S, Chen C-J, Lin Y-C. "Zombie" Outbreak Caused by Synthetic Cannabinoid. N Engl J Med. 2017 Apr 20;376(16):1596-7. doi: 10.1056/NEJMc1701936. No abstract available. PMID 28425277
- [Background] Frank RG, Pollack HA. Addressing the Fentanyl Threat to Public Health. N Engl J Med. 2017 Feb 16;376(7):605-607. doi: 10.1056/NEJMp1615145. No abstract available. PMID 28199808
- [Background] Khaled SM, Hughes E, Bressington D, Zolezzi M, Radwan A, Badnapurkar A, Gray R. The prevalence of novel psychoactive substances (NPS) use in non-clinical populations: a systematic review protocol. Syst Rev. 2016 Nov 21;5(1):195. doi: 10.1186/s13643-016-0375-5. PMID 27871332
- [Background] Kunst LE, Gebhardt WA. Prevalence and Psychosocial Correlates of Party-Drug Use and Associated Problems among University Students in the Netherlands. Subst Use Misuse. 2018 Oct 15;53(12):2077-2088. doi: 10.1080/10826084.2018.1455700. Epub 2018 Apr 18. PMID 29668345
- [Background] Palamar JJ, Barratt MJ, Ferris JA, Winstock AR. Correlates of new psychoactive substance use among a self-selected sample of nightclub attendees in the United States. Am J Addict. 2016 Aug;25(5):400-7. doi: 10.1111/ajad.12403. Epub 2016 Jul 15. PMID 27419383
- [Background] Ridpath A, Driver CR, Nolan ML, Karpati A, Kass D, Paone D, Jakubowski A, Hoffman RS, Nelson LS, Kunins HV; Centers for Disease Control and Prevention (CDC). Illnesses and deaths among persons attending an electronic dance-music festival - New York City, 2013. MMWR Morb Mortal Wkly Rep. 2014 Dec 19;63(50):1195-8. PMID 25522087
- [Background] Fox J, Smith A, Yale A, Chow C, Alaswad E, Cushing T, Monte AA. Drugs of Abuse and Novel Psychoactive Substances at Outdoor Music Festivals in Colorado. Subst Use Misuse. 2018 Jun 7;53(7):1203-1211. doi: 10.1080/10826084.2017.1400067. Epub 2017 Nov 17. PMID 29148866
- [Background] Liakoni E, Dolder PC, Rentsch KM, Liechti ME. Presentations due to acute toxicity of psychoactive substances in an urban emergency department in Switzerland: a case series. BMC Pharmacol Toxicol. 2016 May 26;17(1):25. doi: 10.1186/s40360-016-0068-7. PMID 27228985
- [Background] Palamar JJ, Salomone A, Gerace E, Di Corcia D, Vincenti M, Cleland CM. Hair testing to assess both known and unknown use of drugs amongst ecstasy users in the electronic dance music scene. Int J Drug Policy. 2017 Oct;48:91-98. doi: 10.1016/j.drugpo.2017.07.010. Epub 2017 Aug 12. PMID 28810159
- [Background] Miliano C, Margiani G, Fattore L, De Luca MA. Sales and Advertising Channels of New Psychoactive Substances (NPS): Internet, Social Networks, and Smartphone Apps. Brain Sci. 2018 Jun 29;8(7):123. doi: 10.3390/brainsci8070123. PMID 29966280
- [Background] Robach P, Trebes G, Lasne F, Buisson C, Mechin N, Mazzarino M, de la Torre X, Roustit M, Kerivel P, Botre F, Bouzat P. Drug Use on Mont Blanc: A Study Using Automated Urine Collection. PLoS One. 2016 Jun 2;11(6):e0156786. doi: 10.1371/journal.pone.0156786. eCollection 2016. PMID 27253728
- [Background] Orsini J, Din N, Elahi E, Gomez A, Rajayer S, Malik R, Jean E. Clinical and epidemiological characteristics of patients with acute drug intoxication admitted to ICU. J Community Hosp Intern Med Perspect. 2017 Sep 19;7(4):202-207. doi: 10.1080/20009666.2017.1356189. eCollection 2017 Oct. PMID 29046744
- [Background] Helander A, Backberg M, Hulten P, Al-Saffar Y, Beck O. Detection of new psychoactive substance use among emergency room patients: results from the Swedish STRIDA project. Forensic Sci Int. 2014 Oct;243:23-9. doi: 10.1016/j.forsciint.2014.02.022. Epub 2014 Mar 6. PMID 24726531
- [Background] Spiller HA, Ryan ML, Weston RG, Jansen J. Clinical experience with and analytical confirmation of "bath salts" and "legal highs" (synthetic cathinones) in the United States. Clin Toxicol (Phila). 2011 Jul;49(6):499-505. doi: 10.3109/15563650.2011.590812. PMID 21824061
- [Background] Beck O, Franzen L, Backberg M, Signell P, Helander A. Toxicity evaluation of alpha-pyrrolidinovalerophenone (alpha-PVP): results from intoxication cases within the STRIDA project. Clin Toxicol (Phila). 2016 Aug;54(7):568-75. doi: 10.1080/15563650.2016.1190979. PMID 27412885
- [Background] Backberg M, Beck O, Hulten P, Rosengren-Holmberg J, Helander A. Intoxications of the new psychoactive substance 5-(2-aminopropyl)indole (5-IT): a case series from the Swedish STRIDA project. Clin Toxicol (Phila). 2014 Jul;52(6):618-24. doi: 10.3109/15563650.2014.920088. Epub 2014 Jun 4. PMID 24895941